CLINICAL TRIAL: NCT05418335
Title: Investigation of the Effects of Vitamin D Levels on Oral Health in Stroke Patients
Brief Title: Oral Health and Vitamin D in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Elif yaksi, Medical Doctor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-EY-06
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-06

CONDITIONS: Stroke; Oral Disease; D Vitamin Deficiency
MeSH Terms: conditions — Stroke; Mouth Diseases; Vitamin D Deficiency | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stroke group: stroke history at least 3 months ago
  Interventions: Other: Clinical examination, functional status evaluation
- Control group: Healthy control
  Interventions: Other: Clinical examination, functional status evaluation

INTERVENTIONS:
Other: Clinical examination, functional status evaluation — Barthel Index, Oral Health Impact Profile 14, Beck Depression Inventory, Stroke Impact Scale 3, Plaque Index, Calculus Index, Periodontal Disease Index, Simplified Oral Hygiene Index assesment, DMFT Index

SUMMARY:
Stroke is a common, serious and restrictive global health problem. Restricting the activities of daily living of stroke patients impairs patients' ability to pay attention to oral hygiene. Facial paresis and tongue weakness due to stroke may cause a decrease in the control of dental prostheses and the removal of food residues in the oral cavity. Food residues and saliva contaminated with bacteria as a result of poor oral hygiene can result in pneumonia when aspirated due to oropharyngeal dysphagia. In the literature, it has been shown that there are significant relationships between periodontal health and vitamin D and calcium intake, and that dietary supplementation with calcium and vitamin D can improve periodontal health, increase bone mineral density in the mandible, and inhibit alveolar bone resorption. In line with all these data, our hypothesis in this study is to investigate the relationship between oral health and vitamin D levels in stroke patients in rehabilitation units.

DETAILED DESCRIPTION:
Stroke is a common, serious and restrictive global health problem. In most countries, stroke is among the second or third most common cause of death and is one of the main causes of acquired disability in adults. Although the first attack is usually not fatal in stroke patients, it can often have long-term consequences for patients and their families. Although notable advances have been made in the medical management of stroke, treatment for most stroke patients is based on care and rehabilitation. Motor, perceptual, and cognitive impairments after stroke can have adverse effects on daily functions, reducing health-related quality of life. Restricting the activities of daily living of stroke patients impairs patients' ability to pay attention to oral hygiene. Facial paresis and tongue weakness due to stroke may cause a decrease in the control of dental prostheses and the removal of food residues in the oral cavity. Food residues and saliva contaminated with bacteria as a result of poor oral hygiene can result in pneumonia when aspirated due to oropharyngeal dysphagia.In addition, reduced tongue pressure fails to push the food bolus into the pharynx. Decreased lip strength causes saliva to flow during chewing. Hyposalivation causes a lack of lubrication in the oral mucosa. Abnormal oral sensory function, rapid and improper swallowing of food causes choking and aspiration, and aspiration pneumonia. Incompatible orofacial function leads to low chewing efficiency, limited food selection, and malnutrition. In addition, the risk of poor periodontal health is associated with stroke recurrence and more severe stroke. Third, severe periodontitis, which leads to decreased bite force and increased tooth mobility during chewing, impairs chewing and food intake, affecting oral health conditions.Vitamin D plays a critical role in mediating calcium absorption and regulating musculoskeletal health.There are reports of the benefit of vitamin D and calcium supplementation in the treatment of periodontal disease. Some previous studies reported that calcium and vitamin D supplementation reduced tooth loss and alveolar bone resorption, but could not reach a clear conclusion because of the heterogeneous composition of the study groups or because it did not directly measure periodontal disease status. More recent studies have shown that there are significant associations between periodontal health and the intake of vitamin D and calcium, and that dietary supplementation with calcium and vitamin D can improve periodontal health, increase bone mineral density in the mandible, and inhibit alveolar bone resorption. In line with all these data, our hypothesis in this study is to investigate the relationship between oral health and vitamin D levels in stroke patients in rehabilitation units.

ELIGIBILITY:
Inclusion Criteria:

* Having a history of ischemic stroke at least 3 months
* Age between 50-75

Exclusion Criteria:

* The patient has moderate to severe dementia or mental retardation, which may cause limitations in examination, testing and treatment.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients and healthy control group will be included in the study.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Barthel Index | Baseline
  It is a simple, understandable index that includes all the parameters of daily living activities. It consists of 10 sub-headings: eating, bathing, self-care, dressing, bladder control, bowel control, toilet use, chair/bed transfer, mobility, and use of stairs. Its scoring ranges from 0-100.
Oral Health Impact Profile -14 | Baseline
  Oral health-related quality of life is the individual's personal perception of how oral health affects their quality of life and general health. Oral health impact profile is a scale system that evaluates this perception with two questions on functional limitation, physical pain, psychological discomfort, physical, psychological and social disability and handicap. It is concluded that as the total score increases, the severity of the problem increases and the quality of life decreases.
  It is a scale that evaluates oral health-related quality of life with a questionnaire consisting of a total of 14 questions and 7 sub-headings (functional limitation, physical pain, psychological discomfort, physical, psychological and social disability and disability).
  Each item is scored as 0 (never), 1 (hardly ever), 2 (occasionally), 3 (fairly often), 4 (very often). High score indicates reduced quality of life15.
DMFT Index (Decayed-Missing-Filled-Teeth ) | Baseline
  It shows the number of decayed teeth, filled teeth and teeth extracted due to caries per capita
Periodontal Disease Index | Baseline
  The mesial, distal, facial and lingual areas of each of the teeth are evaluated.

SECONDARY OUTCOMES:
Beck Depression Inventory | Baseline
  It is used to measure physical, emotional and cognitive symptoms such as hopelessness, irritability, guilt, fatigue, and weight loss encountered in depression, was used for evaluation. Scoring in BDI is evaluated progressively from absence of symptoms to severe symptoms. Total score ranged from 0 (no depression) to 63 points (severe depression)
Plaque Index | Baseline
  It is used to evaluate the level and rate of plaque formation on tooth surfaces
Gingival Index | Baseline
  Löe & Silness gingival index values are used to determine gingival inflammation. The mesial, distal, lingual and vestibule gingival conditions of the teeth determined in each sextant are evaluated by scoring between 0-3.Gingival index; grade 0, normal gingiva; grade 1, mild inflammation, slight change in color, slight edema; no bleeding on palpation; grade 2, moderate inflammation, hyperemia, edema, and glazing; bleeding on palpation; grade 3, severe inflammation, marked hyperemia and edema, ulcerations; tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Elif Yakşi, Merkez, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided